CLINICAL TRIAL: NCT03480451
Title: Targeted Intervention for Patient Centered Outcome in Patients With Idiopathic Pulmonary Fibrosis
Acronym: IPF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study considered futile
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Vijaya Ramalingam, Assistant Professor of Medicine, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 28280
Record Dates: First submitted 2016-12-12; First posted 2018-03-29 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): This project is being withdrawn. No revisions to ARM is available.
  Patients will undergo consultation and education by members of a pre-determined multi-disciplinary team that aims to bring a predetermined set of services to the patient in a coordinated and scheduled manner in order to facilitate a comprehensive and through approach to the patient's entire well being
  Interventions: Other: Multi-Disciplinary Patient Centered Rehab and Education

INTERVENTIONS:
Other: Multi-Disciplinary Patient Centered Rehab and Education — This project is being withdrawn. No revisions to Intervention is available.
  Patients will undergo consultation and education by members of a pre-determined multi-disciplinary team that aims to bring a predetermined set of services to the patient in a coordinated and scheduled manner in order to facilitate a comprehensive and through approach to the patient's entire well being

SUMMARY:
Idiopathic pulmonary fibrosis (IPF), a chronic fibrotic lung disease of unknown cause, is characterized by relentless progression, with a three-year mortality of up to 50%. IPF has high morbidity, with 90% of patients reporting dyspnea at the time of diagnosis and this is strongly correlated with quality of life and mortality. As IPF progress, breathlessness worsens, physical functional capacity declines, and health-related quality of life deteriorates. Pulmonary rehabilitation (PR) can improve well-being in patients with other chronic lung disease, but little is known regarding PR in IPF.

DETAILED DESCRIPTION:
The hypothesis is that the provision of a comprehensive pulmonary rehabilitation program to patients with IPF will significantly improve participant health related quality of life. The objective is to develop a comprehensive, multi-disciplinary 12-week PR program with disease specific educational components for IPF patients. The specific aims of the proposal is to evaluate the effect of the comprehensive PR program on 1) improvements in quality of life using the Medical Outcomes Study 36-Item Short Form 36 (SF-36), a quality of life instrument and 2) improvements in patient self-reported dyspnea scores using the chronic respiratory questionnaire. The investigator intends to evaluate sustained benefits of the PR intervention, changes in depression, anxiety, stress and functional physical capacity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF confirmed by lung biopsy or by characteristic pattern on high resolution computed tomogram (HRCT)
* No identifiable cause of lung fibrosis
* PR not received in the past year
* Ability to walk

Exclusion Criteria:

* History of unstable angina
* Deterioration cardiac or neurological disease
* Pregnancy or lactation
* Degenerative arthritis or other limitation to mobility
* PR in the past 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Assess the change in coping skills for patients with IPF before and after a comprehensive pulmonary rehabilitation program. | 12 months
  This project is being withdrawn. No revisions to Outcomes is available. Will use COPE questionnaire.
Assess the change in quality of life for patients with IPF before and after a comprehensive pulmonary rehabilitation program. | 12 months
  Will use 36-item SF questionnaire.
Assess the change in depression, anxiety for patients with IPF before and after a comprehensive pulmonary rehabilitation program. | 12 months
  Will use DASS-21 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Ramalingam, MD, Principal Investigator — Medical College of WI
Locations (1):
- Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Meltzer EB, Noble PW. Idiopathic pulmonary fibrosis. Orphanet J Rare Dis. 2008 Mar 26;3:8. doi: 10.1186/1750-1172-3-8. PMID 18366757
- [Background] Bjoraker JA, Ryu JH, Edwin MK, Myers JL, Tazelaar HD, Schroeder DR, Offord KP. Prognostic significance of histopathologic subsets in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 1998 Jan;157(1):199-203. doi: 10.1164/ajrccm.157.1.9704130. PMID 9445300
- [Background] Swigris JJ, Kuschner WG, Jacobs SS, Wilson SR, Gould MK. Health-related quality of life in patients with idiopathic pulmonary fibrosis: a systematic review. Thorax. 2005 Jul;60(7):588-94. doi: 10.1136/thx.2004.035220. PMID 15994268
- [Background] Olson AL, Brown KK, Swigris JJ. Understanding and optimizing health-related quality of life and physical functional capacity in idiopathic pulmonary fibrosis. Patient Relat Outcome Meas. 2016 May 17;7:29-35. doi: 10.2147/PROM.S74857. eCollection 2016. PMID 27274328
- [Background] Belkin A, Swigris JJ. Health-related quality of life in idiopathic pulmonary fibrosis: where are we now? Curr Opin Pulm Med. 2013 Sep;19(5):474-9. doi: 10.1097/MCP.0b013e328363f479. PMID 23851327
- [Background] Morisset J, Dube BP, Garvey C, Bourbeau J, Collard HR, Swigris JJ, Lee JS. The Unmet Educational Needs of Patients with Interstitial Lung Disease. Setting the Stage for Tailored Pulmonary Rehabilitation. Ann Am Thorac Soc. 2016 Jul;13(7):1026-33. doi: 10.1513/AnnalsATS.201512-836OC. PMID 27064659
- [Background] Lacasse Y, Martin S, Lasserson TJ, Goldstein RS. Meta-analysis of respiratory rehabilitation in chronic obstructive pulmonary disease. A Cochrane systematic review. Eura Medicophys. 2007 Dec;43(4):475-85. PMID 18084170
- [Background] Nici L, ZuWallack R; American Thoracic Society Subcommittee on Integrated Care of the COPD Patient. An official American Thoracic Society workshop report: the Integrated Care of The COPD Patient. Proc Am Thorac Soc. 2012 Mar;9(1):9-18. doi: 10.1513/pats.201201-014ST. PMID 22421582
- [Background] Harrison SL, Greening NJ, Williams JE, Morgan MD, Steiner MC, Singh SJ. Have we underestimated the efficacy of pulmonary rehabilitation in improving mood? Respir Med. 2012 Jun;106(6):838-44. doi: 10.1016/j.rmed.2011.12.003. Epub 2011 Dec 23. PMID 22197576